CLINICAL TRIAL: NCT04833673
Title: The Effects of Relaxation Techniques on Pain, Fatigue and Kinesiophobia in Multiple Sclerosis Patients: A Three Arms Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gülşah Kesik, res.ass., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 333
Record Dates: First submitted 2021-04-05; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2020-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Pain, Chronic; Fatigue Syndrome, Chronic; Kinesiophobia
Keywords: multiple sclerosis; pain; fatigue; kinesiophobia; relaxation techniques; muscle relaxation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Chronic Pain; Fatigue Syndrome, Chronic; Kinesiophobia; Multiple Sclerosis; Pain; Fatigue

STUDY DESIGN:
Intervention Model Description: A Three Arms Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PMR (Experimental): The PMR intervention involving tensing and relaxing the body muscles accompanied with deep breathing. The researchers told each
  participant to sit in a soundless and breathable room and in a comfortable position before each session at their home. The participants performed tensing and relaxing for each body part in order, starting with the facial muscles and head, followed by neck, shoulders, chest, abdomen, legs, and feet; all muscle tension and relaxation procedures were performed with deep breathing. The participants were instructed to tense a specified group of muscles for 5 s and relax it for 10 s while breathing out. Moreover, throughout this exercise, the participants imagined a wave of relaxation flowing over their body.
  Interventions: Behavioral: PMR: Progressive Muscle Relaxation
- BRT (Experimental): Within the scope of this technique, first of all, the participants were asked to focus on a word that relieves them such as love, health or well-being. And so, the participants were asked to be in comfortable position in a silent and breathable room with the closed eyes, relax their muscles from the sole of their feet and progressing up to their face gradually, keep them relaxed, accompanied with deep breathing, be aware of their breathing, exhale gently. They continue these practices for 20 minutes and try to relax their muscles. After finishing the duration, they sit quietly for several minutes with eyes closed and later with eye opened.
  Interventions: Behavioral: BRT:Benson Relaxation Technique
- CG (No Intervention): Regarding CG, the participants were invited to the same room and received only a single time attention-matched education on "Living with MS"; including definition of MS, dietary advices for MS patients. The attention-matched education was performed face to face and lasted for 10 min. All participants in the three study groups also received usual treatment and care.

INTERVENTIONS:
Behavioral: PMR: Progressive Muscle Relaxation — tensing and relaxing the body muscles accompanied with deep breathing
  Arms: PMR
Behavioral: BRT:Benson Relaxation Technique — relaxation using mental imagery and mediation
  Arms: BRT

SUMMARY:
Even though, current treatments including IVIG, corticosteroids, biological agents can provide positive effects on MS symptoms, MS cannot be cured completely today. Therefore, in addition to the available medical treatment options, patients may tend towards complementary and integrative therapies. Relaxation techniques are one of the non-pharmacological and side-effect-free therapy options that are currently used to alleviate the symptoms of many different chronic diseases. Progressive muscle relaxation exercise (PMR) and Benson relaxation technique (BRT) are two common types of relaxation techniques recommended for symptom management in chronic diseases owing to simple to learn and apply compared to other complementary and integrative methods for patients. PMR is uncomplicated and low-cost method, originally designed by Jacobson (1938), which helps individuals to feel calmer through consecutive muscle tension and relaxation of a muscle group. This method can relieve muscle tension, facilitate sleep, and reduce severity of pain and fatigue. There are studies in the literature reporting the positive effects of PMR on fatigue, sleep quality, quality of life, anxiety and stress in MS patients. One of these techniques which is well tolerated is BRT, designed by Herbert Benson in the 1970s as a nonpharmacologic and behavioral method. This technique led to relaxation using mental imagery and mediation. BRT creates a relaxation influence in the body by decreasing the sympathetic nervous system activity and increasing the parasympathetic nervous system activity. There are few studies in the literature reporting that BRT is beneficial on pain and fatigue in MS patients.To the best of our knowledge, there is no study on the impact of relaxation techniques on pain, fatigue and kinesophobia in MS patients. The aim of this study was to examine and compare the effects of PMR and BRT on abovementioned symptoms in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* having relapsing-remitting MS type and not had an attack during the study
* not receiving any other complementary and integrative therapy during the research,
* with an Expanded Disability Status Scale score of 5.5 and below,
* volunteer to participate in study

Exclusion Criteria:

* having physical or mental health problems that can interfere with communication
* having heart failure, COPD, asthma disease, renal failure, musculoskeletal problem such as fracture, plaster cast, amputation, fibromyalgia, ankylosing spondylitis, rheumatoid arthritis, deep anemia (hmg <8 mg / dl) or oncological diagnoses
* not having undergone any surgical operation in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Fatigue | 12 weeks
  Fatigue Severity Scale

SECONDARY OUTCOMES:
Chronic Pain | 12 weeks
  VAS
Kinesiophobia | 12 weeks
  Tampa Scale for Kinesophobia

CONTACTS AND LOCATIONS:
Overall Officials: gulsah kesik, MSc, Principal Investigator — research assisstant
Locations (1):
- Hacettepe University, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Private and personal information of the participants is not open to sharing.

REFERENCES:
- [Derived] Kesik G, Ozdemir L, Mungan Ozturk S. The Effects of Relaxation Techniques on Pain, Fatigue, and Kinesiophobia in Multiple Sclerosis Patients: A 3-Arm Randomized Trial. J Neurosci Nurs. 2022 Apr 1;54(2):86-91. doi: 10.1097/JNN.0000000000000620. PMID 35149625